CLINICAL TRIAL: NCT07064278
Title: Prognostic Significance of Bronchoscopy and CT Score Combined With Monocyte Subsets in Pediatric Patients With Refractory Mycoplasma Pneumoniae Pneumonia
Brief Title: Combined Diagnostic Approach for Refractory Mycoplasma Pneumonia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Hebei Province (Other)
Responsible Party: Principal Investigator, Fangfang Li, Principal Investigator, Children's Hospital of Hebei Province
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-HCH-032
Record Dates: First submitted 2025-06-30; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Refractory Mycoplasma Pneumoniae Pneumonia
Keywords: Pediatric refractory Mycoplasma pneumoniae pneumonia; Bronchoscopy; CT score; Monocyte subpopulation; Prognosis
MeSH Terms: conditions — Pneumonia, Mycoplasma | interventions — Bronchoalveolar Lavage; Azithromycin; Doxycycline; Prednisone; Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Combined Diagnostic and Therapeutic Approach (Experimental): Participants received conventional treatment (supportive care and sequential azithromycin therapy) plus interventions guided by a multi-dimensional assessment. Treatment adjustments were made based on bronchoscopy, CT scoring, and monocyte analysis results. These included: removal of mucous plugs, switching to doxycycline for azithromycin resistance, and adding prednisone for excessive inflammation.
  Interventions: Procedure: Bronchoscopy with Bronchoalveolar Lavage; Procedure: Chest CT with Scoring; Diagnostic Test: Monocyte Subpopulation Analysis; Drug: Azithromycin, Doxycycline, Prednisone
- Control: Conventional Treatment (Active Comparator): Participants received conventional treatment, including supportive care and sequential azithromycin therapy. The regimen consisted of intravenous azithromycin (10 mg/kg/day) for 5 days, followed by a 4-day break and then oral azithromycin for 3 days, repeated for 3 cycles (total duration: 21 days). Supportive care for both groups included antitussives, bronchodilators, and antipyretics as needed.
  Interventions: Drug: Azithromycin, Doxycycline, Prednisone; Other: Supportive Care

INTERVENTIONS:
Procedure: Bronchoscopy with Bronchoalveolar Lavage — Flexible bronchoscopy to assess airway patency, remove mucous plugs, and collect bronchoalveolar lavage (BAL) fluid for microbiological and cytological analysis.
  Arms: Experimental: Combined Diagnostic and Therapeutic Approach
Procedure: Chest CT with Scoring — Chest CT scans at baseline and day 14 to quantitatively assess lesion range, lesion type, pleural effusion, and lymphadenectasis (Total score: 0-13).
  Arms: Experimental: Combined Diagnostic and Therapeutic Approach
Diagnostic Test: Monocyte Subpopulation Analysis — Flow cytometry analysis of peripheral blood to phenotype monocyte subsets (Classical, Intermediate, Non-classical) at baseline and day 14 to guide immunomodulatory therapy.
  Arms: Experimental: Combined Diagnostic and Therapeutic Approach
Drug: Azithromycin, Doxycycline, Prednisone — Sequential azithromycin as baseline therapy. Doxycycline (4 mg/kg/day) was used if BAL results confirmed azithromycin resistance. Oral prednisone (1 mg/kg/day for 5 days) was added if intermediate monocytes were >15%.
Other: Supportive Care — Management of cough, wheezing, and fever based on clinical symptoms.
  Arms: Control: Conventional Treatment

SUMMARY:
This study evaluates whether a combined approach using bronchoscopy, chest CT scoring, and monocyte subpopulation analysis can improve clinical outcomes for children with refractory Mycoplasma pneumoniae pneumonia (RMPP) when compared to conventional treatment. The goal is to determine if this multi-dimensional assessment can lead to more personalized and effective treatment, resulting in shorter recovery times, lower recurrence rates, and better quality of life.

DETAILED DESCRIPTION:
Refractory Mycoplasma pneumoniae pneumonia (RMPP) is a significant clinical challenge in pediatrics, characterized by persistent symptoms despite standard macrolide therapy. This condition often results from a combination of pathogen resistance and excessive host inflammatory responses. Traditional management often fails to adequately assess airway obstruction, quantify lung damage, or characterize the patient's immune status, leading to delayed or suboptimal interventions. This single-center, prospective, randomized controlled trial was designed to address these gaps. A total of 260 children with RMPP were randomly assigned to either an experimental group or a control group. The control group received conventional treatment with sequential azithromycin. The experimental group received conventional treatment plus interventions guided by a multi-dimensional assessment: bronchoscopy with lavage to clear airways and guide antibiotic choice, CT scoring to quantify lung lesion severity and adjust treatment intensity, and monocyte subpopulation analysis to guide immunomodulatory therapy (e.g., corticosteroids). The study hypothesis is that this integrated, personalized approach will significantly improve clinical prognosis, reduce symptom duration and hospitalization, and enhance long-term outcomes compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1-12 years.
* Diagnosed with Mycoplasma pneumoniae pneumonia (MPP) based on clinical symptoms (persistent cough, fever ≥38.5°C for ≥5 days), positive serological tests (IgM antibodies ≥1:160), and chest imaging findings (consolidation or ground-glass opacity).
* Defined as refractory MPP, with no improvement or worsening of symptoms (e.g., fever duration >7 days, increasing respiratory distress) after ≥7 days of standard macrolide therapy.

Exclusion Criteria:

* Presence of severe comorbidities (e.g., congenital heart disease, primary immunodeficiency, chronic lung disease).
* Confirmed bacterial or viral coinfection.
* Known allergies to macrolides or sedatives used for bronchoscopy.
* Guardians refused to provide informed consent.
* Deemed unfit for bronchoscopy (e.g., unstable hemodynamics).

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Time to fever resolution | From date of randomization until the first date of sustained (≥24 hours) temperature <37.5°C, assessed daily for up to 21 days
  Time in days from study enrollment until body temperature is maintained at <37.5°C for at least 24 hours
Time to cough resolution | From date of randomization until the first date of cough frequency ≤10 per day, assessed daily for up to 21 days
  Time in days from study enrollment until cough frequency is ≤10 coughs per day.
Change in CT score | Assessed at baseline and Day 14 post-treatment
  The change in the total chest CT score from baseline to 14 days post-treatment. The score assesses lesion range, lesion type, pleural effusion, and lymphadenectasis. The score ranges from 0-13, where a lower score indicates less severe lung involvement; thus, a greater reduction in the score indicates a better outcome.
Change in serum Tumor Necrosis Factor-alpha (TNF-α) level | Assessed at baseline and Day 14 post-treatment
  Change in serum TNF-α level from baseline to post-treatment.
Change in serum Interleukin-6 (IL-6) level | Assessed at baseline and Day 14 post-treatment
  Change in serum IL-6 level from baseline to post-treatment.
Change in serum C-reactive protein (CRP) level | Assessed at baseline and Day 14 post-treatment
  Change in serum CRP level from baseline to post-treatment.

SECONDARY OUTCOMES:
Duration of hospitalization | From date of hospital admission until date of hospital discharge, assessed up to 21 days
  Total length of stay in the hospital, measured in days.
Duration of ICU stay | From date of ICU admission until date of ICU discharge, assessed up to 21 days
  Total length of stay in the Intensive Care Unit (ICU), measured in days.
6-month recurrence rate | Assessed at 6 months post-discharge
  Percentage of patients re-admitted for Mycoplasma pneumoniae pneumonia with positive IgM serology within 6 months of discharge.
Quality of life score | Assessed at 6 months post-discharge
  Assessed using the Pediatric Quality of Life Inventory (PedsQL 4.0) Generic Core Scales. The questionnaire assesses physical, emotional, social, and school functioning. Scores are transformed to a 0-100 scale, where 0 is the minimum value and 100 is the maximum value. A higher score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Children's Hospital, Shijiazhuang, Hebei, China